CLINICAL TRIAL: NCT02100449
Title: Role of Lung Ultrasound Imaging and Pulsed-wave Doppler in the Assessment of Lung Consolidations in Mechanically Ventilated Patients.
Brief Title: Role of Lung Ultrasound and Pulsed-wave Doppler in Lung Consolidations in Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14.005
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Atelectasis; Pneumonia
Keywords: Atelectasis; Pneumonia; Lung ultrasound; Doppler
MeSH Terms: conditions — Pulmonary Atelectasis; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung ultrasound and Doppler, pneumonia (Other): In this group, a lung ultrasound examination using pulsed-wave Doppler will be performed in patients with high clinical suspicion of pneumonia on Day 0. A bronchoalveolar lavage will also be performed on Day 0.
  Interventions: Other: Lung ultrasound and Doppler (Day 0)
- Lung ultrasound and Doppler, atelectasis (Other): Patients without clinically active pulmonary disease but presenting a consolidation of suspected atelectatic nature. Fever, hypothermia, leucocytosis and leucopenia will not be present. Tracheal secretions will remain unchanged. There will be no deterioration of oxygenation. In this group, a lung ultrasound examination using pulsed-wave Doppler will be performed on Day 0.
  Interventions: Other: Lung ultrasound and Doppler (Day 0)

INTERVENTIONS:
Other: Lung ultrasound and Doppler (Day 0) — In patients presenting a consolidation of suspected atelectatic nature, a lung ultrasound examination using pulsed-wave Doppler will be performed on Day 0.
  Arms: Lung ultrasound and Doppler, atelectasis
Other: Lung ultrasound and Doppler (Day 0) — In patients presenting a consolidation of suspected infectious nature, a lung ultrasound examination using pulsed-wave Doppler will be performed on Day 0. A bronchoalveolar lavage will also be performed on Day 0.
  Arms: Lung ultrasound and Doppler, pneumonia

SUMMARY:
In infectious lung consolidations, the inhibition of hypoxic pulmonary vasoconstriction (HPV) results in a higher regional acceleration time (RAcT) compared to the RAcT measured in atelectatic consolidations.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia has a considerable impact on morbidity and mortality in intensive-care patients. Chest radiography, which is the most frequently used imagery test for bedside lung evaluation in mechanically ventilated patients, is recognized to be poorly sensitive and non-specific for the diagnosis of ventilator-associated pneumonia. Bronchoalveolar lavage using a bronchoscope remains the most reliable tool for the diagnosis of this nosocomial infection. However, a bronchoscopy may not be feasible in all patients and waiting time before final results become available may cause a delay in the initiation of the treatment, thus increasing the risk of mortality. Lung ultrasound is a promising non-invasive, non-radiant, portable and easy to use tool especially in critically-ill patients.

Dependent atelectasis is a frequent phenomenon in mechanically ventilated patients. The presence of clinical infection signs raises the question of the nature of the infiltrate. A consolidation of infectious nature differs from atelectasis by its local hypoxic pulmonary vasoconstriction inhibition. In patients breathing spontaneously, it is possible to detect this difference using the RAcT, measured by pulsed-wave Doppler in an arterial blood vessel located in a pulmonary consolidation visible by ultrasound examination. The use of pulsed-wave Doppler to measure the RAcT in a consolidation added to the value of general lung ultrasound could help determine the infectious or atelectatic nature of a consolidation in mechanically ventilated patients. However, the RAcT has never been studied in patients under positive pressure ventilation. In this observational study, the investigators will explore the role of measuring the RAcT and of general lung ultrasound as a diagnostic tool to detect pneumonia in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Under mechanical ventilation and presenting one or more consolidations on chest radiography or CT scan

Exclusion Criteria:

* Participation to another study
* Poor echogenicity (morbid obesity, multiple thoracic dressings)
* Contra-indications to superior limbs or torso mobilization
* Contra-indications to bronchoscopy
* Antibiotics initiated more than 24 hours but less than 72 hours before inclusion or changes in the antibiotic regimen in the last 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-06-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
RAcT in lung consolidations | During lung ultrasound examination - Day 0
  Regional acceleration time measured by lung ultrasound and pulsed-wave Doppler

SECONDARY OUTCOMES:
Presence of visible blood vessels on colour Doppler in lung consolidations | During lung ultrasound examination - Day 0
  Graded semi-quantitatively (absence, single, multiple branching)
Presence of dynamic air bronchograms in lung consolidations | During lung ultrasound examination - Day 0
  To-and-fro respiratory movement of punctiform or linear hyperechoic artifacts (absence or presence)
Presence of sub-pleural consolidations | During lung ultrasound examination - Day 0
  Subpleural hypoechoic area with ragged margins (absence or presence)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada